CLINICAL TRIAL: NCT01138280
Title: Effect of Heat Disinfection of HD Water Treatment System on Cardiovascular Events and Outcome in Hemodialysis Patients
Brief Title: Heat Disinfection of HD Water Treatment System in Hemodialysis Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: DER-CHERNG TARNG, Taipei Veterans General Hospital, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VGHIRB 96-12-21A; VGHUST97-P1-01 (Other Grant/Funding Number: Taipei Veterans General Hospital, Taiwan)
Record Dates: First submitted 2010-05-25; First posted 2010-06-07 (Estimated); Last update posted 2010-06-07 (Estimated); Status verified 2005-01

CONDITIONS: All Cause Mortality
Keywords: biofilm formation; proinflammatory cytokines; high sensitive c reactive protein; cardiovascular events; overall mortality; hemodialysis
MeSH Terms: interventions — Kidneys, Artificial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Heat disinfection (Experimental): Experimental arm: Heat disinfection link to RO water treatment system and piping system to dialysis machine
  Interventions: Device: CWP 103H (Gambro, Sweden): a heat disinfection device
- Conventional RO water treatment (No Intervention): Placebo arm: conventional chemical disinfection link to RO water treatment system.

INTERVENTIONS:
Device: CWP 103H (Gambro, Sweden): a heat disinfection device — Heat disinfection can increase temperature to 95c in the RO water treatment system and then in the piping system link to dialysis machines in each hemodialysis center per night
  Other Names: Heat disinfection (temperature up to 95 c); RO water treatment system; piping system; dialysis machine
  Arms: Heat disinfection

SUMMARY:
Hemodialysis (HD) may lead to increase inflammatory response through a number of mechanisms. HD-related inflammation is mainly due to underlying kidney disease, coexisting comorbidities, uremia per se, dialyzer membrane biocompatibility and contaminated dialysis fluid. Accordingly, HD patients are chronically exposed to microinflammation as a result of blood-membrane interaction and dialysis fluid contamination. Among these factors, biofilm formation and contaminated dialysis fluid are closely related to enhanced immune activation in HD patients. Furthermore, only dialysis fluid quality is controllable and preventable. Therefore, to reduce the cardiovascular (CV) events and improve the outcome, it prompts us to conduct a prospective randomized controlled study to explore whether heat disinfection link in HD water treatment system can effectively prevent biofilm formation, to ensure the dialysis fluid purity, and subsequently to improve the patient outcome, in terms of CV events and mortality.

DETAILED DESCRIPTION:
Inflammation is common in individuals with both chronic kidney disease (CKD) and hemodialysis (HD). HD may lead to increased inflammatory response through a number of mechanisms; some of these factors also result in pro-inflammatory cytokine release and consequently cause the overlap between anemia, accelerated atherosclerosis and inflammation. HD-related inflammation is mainly due to underlying kidney disease, coexisting comorbidities, uremia per se, dialyzer membrane biocompatibility and contaminated dialysis fluid. Accordingly, HD patients are chronically exposed to microinflammation as a result of blood-membrane interaction and dialysis fluid contamination. Among these factors, biofilm formation and contaminated dialysis fluid are closely related to enhanced immune activation in HD patients. Furthermore, only dialysis fluid quality is controllable and preventable. Therefore, to correct rHuEPO poor response and reduce the cardiovascular (CV) events, it prompts us to conduct a prospective randomized controlled study to explore as to whether heat disinfection link in HD water treatment system can effectively prevent biofilm formation, to ensure the dialysis fluid purity, and subsequently to improve the patient outcome, in terms of CV events and mortality.

ELIGIBILITY:
Inclusion Criteria:

* age over 20 years and duration of HD over 3 months, and clinically stable

Exclusion Criteria:

* patients with acute infection, malignancy, active autoimmune disease, GI bleeding or blood loss; systemic inflammatory disease; life expectancy less than 3 months, and unwilling to participate in this study.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Actual)
Dates: Start 2005-03; Primary Completion 2009-12 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
CV events, CV | 5 years
all-cause mortality | 5 years

SECONDARY OUTCOMES:
biofilm formation | 5 years
endotoxin level of dialysis water | 5 years
pro-inflammatory cytokine levels in serum | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Der-Cherng Tarng, MD, PhD, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan